CLINICAL TRIAL: NCT00362180
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of Apolipoprotein B(ApoB) Reduction by ISIS 301012 on Liver Triglyceride Content in Subjects With Varying Degrees of Hyperlipidemia
Brief Title: Measure Liver Fat Content After ISIS 301012 (Mipomersen) Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kastle Therapeutics, LLC (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301012-CS10; 2005-005783-90 (EudraCT Number)
Record Dates: First submitted 2006-08-07; First posted 2006-08-09 (Estimated); Results first posted 2015-06-24 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-09

CONDITIONS: Lipid Metabolism, Inborn Errors; Hyperlipidemias; Metabolic Diseases; Hypolipoproteinemia; Hypolipoproteinemias; Hypobetalipoproteinemias; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Congenital Abnormalities; Metabolic Disorder; Hypercholesterolemia; Dyslipidemias; Lipid Metabolism Disorders
Keywords: LDL-cholesterol; apoB-100; apoB-48; triglyceride; HeFH; FHBL
MeSH Terms: conditions — Lipid Metabolism, Inborn Errors; Hyperlipidemias; Metabolic Diseases; Hypolipoproteinemias; Hypobetalipoproteinemias; Metabolism, Inborn Errors; Genetic Diseases, Inborn; Infant, Newborn, Diseases; Congenital Abnormalities; Hypercholesterolemia; Dyslipidemias; Lipid Metabolism Disorders | interventions — mipomersen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- Cohort A: mipomersen (Experimental): Healthy volunteers treated with 6 injections of mipomersen 200 mg over the course of 4 weeks. Injections were given subcutaneously (sc) on days 1, 4, 8, 11, 15 and 22.
  Interventions: Drug: mipomersen
- Cohort A: placebo (Placebo Comparator): Healthy volunteers treated with 6 injections of placebo over the course of 4 weeks. Injections were given subcutaneously (sc) on days 1, 4, 8, 11, 15 and 22.
  Interventions: Drug: Placebo
- Cohort D: mipomersen (Experimental): Participants with impaired fasting glucose and mixed dyslipidemia who were treated with 6 injections of mipomersen 200 mg over the course of 4 weeks. Injections were given subcutaneously (sc) on days 1, 4, 8, 11, 15 and 22.
  Interventions: Drug: mipomersen
- Cohort D: placebo (Placebo Comparator): Participants with impaired fasting glucose and mixed dyslipidemia who were treated with 6 injections of placebo over the course of 4 weeks. Injections were given subcutaneously (sc) on days 1, 4, 8, 11, 15 and 22.
  Interventions: Drug: Placebo
- Cohort E: mipomersen (Experimental): Participants with uncomplicated heterozygous familial hypercholesterolemia (HeFH) treated with weekly mipomersen 200 mg injections for 13 weeks.
  Interventions: Drug: mipomersen
- Cohort E: placebo (Placebo Comparator): Participants with uncomplicated heterozygous familial hypercholesterolemia (HeFH) treated with weekly placebo injections for 13 weeks.
  Interventions: Drug: Placebo
- Cohort F: no intervention (No Intervention): A reference group of participants with familial hypobetalipoproteinemia (FBHL) who did not receive a study intervention. Data gathered for 15 weeks.
- Cohort G: mipomersen (Experimental): Participants with well-controlled Type 2 diabetes mellitus, hypercholesterolemia, and normal triglyceride levels were treated with mipomersen 200 mg weekly for 26 weeks, followed by open-label mipomersen 200 mg weekly for an additional 26 weeks.
  Interventions: Drug: mipomersen
- Cohort G: placebo followed by mipomersen (Placebo Comparator): Participants with well-controlled Type 2 diabetes mellitus, hypercholesterolemia, and normal triglyceride levels were treated with placebo weekly for 26 weeks, followed by open-label mipomersen 200 mg weekly for an additional 26 weeks.
  Interventions: Drug: mipomersen; Drug: Placebo

INTERVENTIONS:
Drug: mipomersen — 200 mg subcutaneous injections
  Other Names: ISIS 301012; mipomersen sodium; Kynamro™
  Arms: Cohort A: mipomersen; Cohort D: mipomersen; Cohort E: mipomersen; Cohort G: mipomersen; Cohort G: placebo followed by mipomersen
Drug: Placebo — subcutaneous injections
  Arms: Cohort A: placebo; Cohort D: placebo; Cohort E: placebo; Cohort G: placebo followed by mipomersen

SUMMARY:
This study will assess what, if any, effect that ISIS 301012 (mipomersen) has on liver triglyceride content in multiple groups of subjects with varying degrees of risk for hepatic steatosis. In order to enroll subject groups with varying degrees of risk, the study has included multiple cohorts (Cohorts A-G). Additions and removal of cohorts has been accomplished with protocol amendments.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled study to measure the effect of treatment with mipomersen on liver triglyceride (TG) content in patients with varying degrees of hyperlipidemia and risk for hepatic steatosis.

The original study design included 4 cohorts (Cohorts A through D). Subsequent protocol amendments added 3 cohorts (Cohorts E, F, and G) to the study, truncated the enrollment of Cohort D, and eliminated Cohorts B and C. The study consisted of up to a 3-week screening period; a 4-week (Cohorts A and D), 13-week (Cohort E), or 52-week (Cohort G) treatment period; and a 20-week post-treatment follow-up period. Cohort F was an observational cohort, and therefore, was not treated with study drug. Patients in this cohort underwent a 15-week Magnetic resonance spectroscopy (MRS) and ultrasound evaluation period.

The study cohorts are:

Cohort A: Healthy volunteers with LDL-C <140 mg/dL (3.6 mmol/L), serum TG <200 mg/dL (2.3 mmol/L), hemoglobin A1c (HbA1c) <6.0%, and hepatic TG content <5% (as measured by MRS at screening). Patients were randomized to mipomersen 200 mg or placebo and treated for 4 weeks.

Cohorts B+C were eliminated in a protocol amendment prior to enrolling any patients and are not discussed further.

Cohort D: In an amendment to the protocol, Cohort D was closed to enrollment. One patient had already been enrolled in the study prior to the amendment. The patient enrolled in this cohort had impaired fasting glucose (defined as fasting blood glucose >6 mmol/L and <7 mmol/L) and mixed dyslipidemia (LDL-C <215 mg/dL [5.6 mmol/L] and serum TG >200 mg/dL [2.3 mmol/L]). The patient was treated with mipomersen 200 mg for 4 weeks.

Cohort E: Patients with uncomplicated heterozygous familial hypercholesterolemia (HeFH) (Alanine aminotransferase (ALT) ≤1.5 * upper limit of normal Upper limit of normal (ULN), no evidence of insulin resistance or metabolic syndrome, and hepatic TG content <5% by MRS at screening). Patients were to remain on their baseline statin ± ezetimibe regimen but were to wash out from other lipid-lowering agents (e.g., fenofibrate, non-dietary omega-3 fatty acids, and niacin) at least 8 weeks prior to the MRS at screening. Patients were randomized to either mipomersen 200 mg or placebo for 13 weeks.

Cohort F: Patients with familial hypobetalipoproteinemia (FHBL) (a documented APOB gene mutation that results in the expression of a truncated form of apo B). Patients in this cohort were evaluated by MRS, ultrasound, and laboratory tests; however, they were not treated with mipomersen or placebo.

Cohort G: Patients with well-controlled type 2 diabetes mellitus (HbA1c ≤8.0%), hypercholesterolemia (LDL-C >100 mg/dL (2.59 mmol/L), and normal serum TG levels (≤200 mg/dL [2.26 mmol/L]). Patients were to have been on a stable dose of antidiabetic and lipid-lowering medications >3 months prior to screening and were expected to remain stable for the duration of the study. Patients were randomized to either mipomersen 200 mg or placebo for 26 weeks, followed by 26 additional weeks of mipomersen 200 mg. Recruiting difficulties caused this cohort to close early.

ELIGIBILITY:
Inclusion Criteria:

* Group A - are healthy subjects
* Group D - has impaired fasting glucose and mixed dyslipidemia
* Group E - has a diagnosis of Heterozygous Familial Hypercholesterolemia (HeFH) and on stable lipid-lowering therapy for 3 months
* Group F - has a diagnosis of Familial Hypobetalipoproteinemia (FHBL)
* Group G - has a diagnosis of Diabetes and hypercholesterolemia

Exclusion Criteria:

* Medical, surgical, laboratory or other conditions which in the judgment of the Physician Investigator would make the subject unsuitable for enrollment, or potentially interfere with subject participation or completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- Amsterdam, Netherlands

REFERENCES:
- [Result] Visser ME, Akdim F, Tribble DL, Nederveen AJ, Kwoh TJ, Kastelein JJ, Trip MD, Stroes ES. Effect of apolipoprotein-B synthesis inhibition on liver triglyceride content in patients with familial hypercholesterolemia. J Lipid Res. 2010 May;51(5):1057-62. doi: 10.1194/jlr.M002915. Epub 2009 Dec 14. PMID 20008831

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Mipomersen: Healthy volunteers treated with 6 injections of mipomersen 200 mg over the course of 4 weeks.
- Cohort A: Placebo: Healthy volunteers treated with 6 injections of placebo over the course of 4 weeks.
- Cohort D: Mipomersen: Participants with impaired fasting glucose and mixed dyslipidemia who were treated with 6 injections of mipomersen 200 mg over the course of 4 weeks.
- Cohort D: Placebo: Participants with impaired fasting glucose and mixed dyslipidemia who were treated with 6 injections of placebo over the course of 4 weeks.
- Cohort F: no Study Intervention: A reference group of participants with familial hypobetalipoproteinemia (FBHL) who did not receive a study intervention. Data gathered for 15 weeks.
Period: Treated Period
Arm/Group | Cohort A: Mipomersen | Cohort A: Placebo | Cohort D: Mipomersen | Cohort D: Placebo | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: no Study Intervention | Cohort G: Mipomersen | Cohort G: Placebo Followed by Mipomersen
Started | 4 | 2 | 1 | 0 | 11 | 10 | 6 | 3 | 1
Completed | 3 | 2 | 1 | 0 | 11 | 9 | 6 | 2 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Period: 20 Week Safety Follow-up
Arm/Group | Cohort A: Mipomersen | Cohort A: Placebo | Cohort D: Mipomersen | Cohort D: Placebo | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: no Study Intervention | Cohort G: Mipomersen | Cohort G: Placebo Followed by Mipomersen
Started | 3 | 2 | 1 | 0 | 11 | 9 | 0 (This observational cohort did not include a safety follow-up period.) | 3 | 1
Completed | 3 | 2 | 1 | 0 | 11 | 9 | 0 | 3 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Mipomersen | Cohort A: Placebo | Cohort D: Mipomersen | Cohort D: Placebo | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: no Study Intervention | Cohort G: Mipomersen | Cohort G: Placebo Followed by Mipomersen | Total
Number analyzed (Participants) | 4 | 2 | 1 | 0 | 11 | 10 | 6 | 3 | 1 | 38
Age, Continuous [Median (Full Range); unit: years] | 58.5 [57 to 65] | 40.5 [24 to 57] | 59.0 [59 to 59] |  | 46.0 [28 to 59] | 50.0 [23 to 63] | 49.5 [29 to 71] | 62.0 [49 to 64] | 58.0 [58 to 58] | 53.5 [23 to 71]
Gender [Number; unit: participants]
  Female | 2 | 1 | 1 |  | 8 | 4 | 1 | 2 | 1 | 20
  Male | 2 | 1 | 0 |  | 3 | 6 | 5 | 1 | 0 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 4 | 1 | 1 |  | 11 | 10 | 6 | 3 | 1 | 37
  Black or African American | 0 | 1 | 0 |  | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Liver Triglyceride (TG) Content As Measured by Magnetic Resonance Spectroscopy (MRS)
Description: Localized proton MRS was used to quantify liver TG concentration. All MRS imaging of the liver was performed using the same 1.5T scanner. The instructions were to cover the entire liver (from just above the dome to just below the inferior tip) using a qualified imaging technique (Yokoo, 2009, Radiology). Liver fat quantification was performed by determining the liver fat fraction (%) derived from MRS using selected Regions of Interest (ROI). The analyst typically looked for the branching of the right portal vein and mapped slices from one scan to the next. There were typically 2 ROIs in the right lobe and 1 in the left lobe. Magnetic resonance spectroscopy imaging ROIs between different scans were selected using anatomical landmarks for both time points.
Time Frame: Baseline, Day 26, Day 99
Population: Full analysis set. In Cohort E: Placebo, Day 99 N=11 instead of 10 because participant did not have a post treatment MRS by Day 26.
Measure: Median (Full Range); unit: percentage of total liver content
Groups:
- Cohort D: Participants with impaired fasting glucose and mixed dyslipidemia who were treated with 6 injections of mipomersen 200 mg over the course of 4 weeks.
- Cohort F: no Study Intervention: Participants with a diagnosis of Familial Hypobetalipoproteinemia (FHBL) and were not treated with mipomersen or placebo.
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: no Study Intervention | Cohort G: Placebo Followed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 11 | 10 | 6 | 1 | 3
percentage of total liver content
  Baseline (Cohort E: Placebo n=11) | 0.2 [0.1 to 0.3] | 1.2 [0.5 to 1.8] | 6.4 [6.4 to 6.4] | 0.8 [0.2 to 3.2] | 1.1 [0.3 to 3.8] | 21.4 [13.2 to 30.1] | 2.6 [2.6 to 2.6] | 2.5 [1.7 to 3.2]
  Day 26 (Cohort E: Placebo n=10) | 0.3 [0.0 to 0.6] | 0.3 [0.0 to 0.5] | 4.45 [4.45 to 4.45] | 0.1 [-0.4 to 0.8] | 0.1 [-2.5 to 0.5] | -1.2 [-2.6 to 4.3] | NA [NA to NA] — Liver TG not collected at day 26 as per protocol | NA [NA to NA] — Liver TG not collected at day 26 as per protocol
  Day 99 (Cohort E: Placebo n=11) | NA [NA to NA] — Liver TG not collected at day 99 as per protocol | NA [NA to NA] — Liver TG not collected at day 99 as per protocol | NA [NA to NA] — Only 1 patient was enrolled in cohort D, there was no day 99 visit for cohort D | -0.0 [-1.5 to 1.3] | 0.4 [-1.7 to 5.1] | 0.8 [-2.0 to 4.3] | -1.0 [-1.0 to -1.0] | 7.8 [1.1 to 14.5]
Statistical Analysis 1: Comparison: Cohort E: Placebo vs Cohort E: Mipomersen; The p-value is a comparison between the placebo group and the mipomersen group in Cohort E as a change from Baseline to Day 26; Test type: Superiority or Other; p = 0.7244, exact Wilcoxon Rank-sum test
Statistical Analysis 2: Comparison: Cohort E: Placebo vs Cohort E: Mipomersen; The p-value is a comparison between the placebo group and the mipomersen group in Cohort E as a change from Baseline to Day 99; Test type: Superiority or Other; p = 0.0513, exact Wilcoxon Rank-sum test

2. Secondary Outcome: Baseline Apolipoprotein B
Description: Samples were taken following an overnight fast.
Time Frame: Baseline
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/wk
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: no Study Intervention | Cohort G: Placebo Followed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 11 | 10 | 6 | 1 | 3
mg/wk | 86 [70 to 102] | 100.5 [76.5 to 102.0] | 155 [155 to 155] | 122.0 [106.0 to 148.0] | 126.5 [109.0 to 153.0] | 31.5 [28.0 to 41.0] | 120.0 [120.0 to 120.0] | 113.0 [90.0 to 132.0]

3. Secondary Outcome: Percent Change in Apolipoprotein B From Baseline to Day 99
Description: Samples were taken following an overnight fast.
Time Frame: Day 26 and Day 99
Population: Full analysis set with last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: No Study Intervention | Cohort G: Placebo Followed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 11 | 10 | 6 | 1 | 3
percent change
  Day 26 | -3.3 [-8.6 to 2.0] | -20.8 [-24.8 to -13.6] | -41.6149 [-41.6149 to -41.6149] | -1.1 [-1.8 to 0.0] | -1.8 [-16.3 to 13.4] | 3.6 [-4.9 to 14.3] | NA [NA to NA] — Apolipoprotein B was not collected at day 26 as per protocol | NA [NA to NA] — Apolipoprotein B was not collected at day 26 as per protocol
  Day 99 | NA [NA to NA] — Apolipoprotein B was not collected at day 99 as per protocol | NA [NA to NA] — Apolipoprotein B was not collected at day 99 as per protocol | NA [NA to NA] — Only 1 patient was enrolled in cohort D, there was no day 99 visit for cohort D | 6.0 [-2.7 to 15.3] | -16.3 [-29.3 to -5.6] | 4.1 [0.0 to 5.9] | -25.8 [-25.8 to -25.8] | -44.2 [-55.6 to -18.2]

4. Secondary Outcome: Baseline Low-Density Lipoprotein Cholesterol
Description: Samples were taken following overnight fast.
Time Frame: Baseline
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/wk
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: No Study Intervention | Cohort G: Placebo Followed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 11 | 10 | 6 | 1 | 3
mg/wk | 103.5 [77.0 to 130.0] | 126.0 [93.0 to 139.5] | 156.0 [156.0 to 156.0] | 148.0 [131.0 to 182.0] | 151.5 [127.0 to 161.0] | 41.5 [37.0 to 55.0] | 147.0 [147.0 to 147.0] | 121.0 [94.0 to 131.0]

5. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol From Baseline to Day 99
Description: Samples were taken following an overnight fast.
Time Frame: Day 26 and Day 99
Population: Full analysis set with last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Cohort G: Placebo Follwed by Mipomersen: Participants with well-controlled Type 2 diabetes mellitus, hypercholesterolemia, and normal triglyceride levels were treated with placebo weekly for 26 weeks, followed by open-label mipomersen 200 mg weekly for an additional 26 weeks.
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D: Mipomersen | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: No Study Intervention | Cohort G: Placebo Follwed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 11 | 10 | 6 | 1 | 3
percent change
  Day 26 | 1.1 [-11.7 to 13.8] | -14.3 [-20.5 to -6.0] | -41.7143 [-41.7143 to -41.7143] | -2.7 [-5.0 to 2.4] | -5.4 [-20.9 to 11.4] | 0.0 [-4.9 to 8.0] | NA [NA to NA] — Low-density lipoprotein was not collected at day 26 as per protocol | NA [NA to NA] — Low-density lipoprotein was not collected at day 26 as per protocol
  Day 99 | NA [NA to NA] — Low-density lipoprotein was not collected at day 99 as per protocol | NA [NA to NA] — Low-density lipoprotein was not collected at day 99 as per protocol | NA [NA to NA] — Only 1 patient was enrolled in cohort D, there was no day 99 visit for cohort D | 0.7 [-9.8 to 13.5] | -15.9 [-36.1 to -12.4] | 2.6 [-5.1 to 9.0] | -19.0 [-19.0 to -19.0] | -33.9 [-63.8 to -18.3]

6. Secondary Outcome: Baseline Total Cholesterol
Description: Samples were taken following an overnight fast.
Time Frame: Baseline
Population: Full analysis set
Measure: Median (Inter-Quartile Range); unit: mg/wk
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D | Cohort E: Placebo | Cohort E: Mipomersen | Cohort F: No Study Intervention | Cohort G: Placebo Followed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 11 | 10 | 6 | 1 | 3
mg/wk | 201.0 [165.0 to 237.0] | 207.0 [176.0 to 213.0] | 263.0 [263.0 to 263.0] | 208.0 [191.0 to 245.0] | 220.5 [189.0 to 248.0] | 107.0 [93.0 to 115.0] | 231.0 [231.0 to 231.0] | 199.0 [171.0 to 208.0]

7. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 99
Description: Samples were taken following an overnight fast.
Time Frame: Day 26 and Day 99
Population: Full analysis set with last observation carried forward.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Cohort A: Placebo | Cohort A: Mipomersen | Cohort D: Mipomersen | Cohort E: Mipomersen | Cohort E: Placebo | Cohort F: No Study Intervention | Cohort G: Placebo Follwed by Mipomersen | Cohort G: Mipomersen
Number analyzed (Participants) | 2 | 4 | 1 | 10 | 11 | 6 | 1 | 3
percent change
  Day 26 | -3.5 [-7.9 to 0.8] | -11.7 [-12.5 to -0.7] | -29.5374 [-29.5374 to -29.5374] | -3.1 [-16.9 to 10.1] | 0.1 [-2.1 to 3.0] | 1.4 [0.0 to 2.7] | NA [NA to NA] — Total cholesterol was not collected at day 26 as per protocol | NA [NA to NA] — Total cholesterol was not collected at day 26 as per protocol
  Day 99 | NA [NA to NA] — Total cholesterol was not collected at day 99 as per protocol | NA [NA to NA] — Total cholesterol was not collected at day 99 as per protocol | NA [NA to NA] — Only 1 patient was enrolled in cohort D, there was no day 99 visit for cohort D | -11.8 [-24.2 to -9.7] | -0.8 [-8.9 to 12.7] | -0.4 [-6.9 to 4.3] | -21.6 [-33.9 to -14.1] | -21.6 [-33.9 to -14.1]

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Placebo: Placebo
- Mipomersen: Mipomersen
- Not Treated: Not Treated
Arm/Group | Placebo | Mipomersen | Not Treated
Serious Adverse Events (participants affected / at risk) | 0/14 | 1/19 | 0/6
Other Adverse Events (participants affected / at risk) | 14/14 | 19/19 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Mipomersen (N=19) | Not Treated (N=6)
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Mipomersen (N=19) | Not Treated (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Eustachian tube disorder (Ear and labyrinth disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2 | 1
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Chest discomfort (General disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 2 | 0
Feeling cold (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 2 | 9 | 0
Injection site discolouration (General disorders) | 0 | 4 | 0
Injection site discomfort (General disorders) | 0 | 5 | 0
Injection site erythema (General disorders) | 0 | 8 | 0
Injection site haematoma (General disorders) | 0 | 4 | 0
Injection site induration (General disorders) | 0 | 3 | 0
Injection site inflammation (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 9 | 0
Injection site pallor (General disorders) | 0 | 2 | 0
Injection site pruritus (General disorders) | 0 | 3 | 0
Injection site reaction (General disorders) | 8 | 10 | 0
Injection site swelling (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 4 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 4 | 0
Nasopharyngitis (Infections and infestations) | 5 | 7 | 1
Pertussis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 4 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 5 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Listless (Psychiatric disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0
Urine abnormality (Renal and urinary disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The limitations to this study are 1) post-hoc amendments that caused early termination of cohorts and limited the accomplishment of study objectives and 2) post-hoc amendments which added cohorts into the study that were not previously specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI gives Sponsor a draft 90 days before publication. Sponsor has the right to demand that confidential information be removed, and can defer publication another 180 days upon notifying PI that it will file a patent application on inventions contained in the draft.